CLINICAL TRIAL: NCT03453112
Title: A 12-week, Multicenter, Randomized, Double-blind, Double-dummy, 2-arm Parallel Group Study Comparing the Efficacy and Safety of Foster 100/6mg NEXThaler, 2 Inhalations b.i.d, Versus Foster 100/6mg pMDI, 2 Puffs b.i.d in Patients With Controlled Asthma
Brief Title: Foster 100/6 mg NEXThaler Versus Foster 100/6mg Pressurized Metered-dose Inhaler (pMDI) in Patients With Controlled Asthma.
Acronym: FORTUNE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-01535BA0-01
Record Dates: First submitted 2018-02-12; First posted 2018-03-05 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Asthma
Keywords: Peek Expiratory Flow (PEF) Lung function tests
MeSH Terms: conditions — Asthma | interventions — Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foster 100/6mg NEXThaler (Experimental): Fixed combination of beclomethasone dipropionate 100mg plus formoterol fumarate 6mg per actuation as inhalation powder with a new dry powder inhaler (NEXThaler)
  Interventions: Drug: Foster 100/6mg NEXThaler
- Foster 100/6mg pMDI (Active Comparator): Fixed combination of beclomethasone dipropionate 100mg plus formoterol fumarate 6mg per actuation as pMDI with Hydrofluoroalkane ( HFA) -134a propellant.
  Interventions: Drug: Foster 100/6mg pMDI

INTERVENTIONS:
Drug: Foster 100/6mg NEXThaler — Fixed combination of beclomethasone dipropionate 100mg plus formoterol fumarate 6mg per actuation as inhalation powder with a new dry powder inhaler
  Arms: Foster 100/6mg NEXThaler
Drug: Foster 100/6mg pMDI — Fixed combination of beclomethasone dipropionate 100mg plus formoterol fumarate 6mg per actuation as pMDI with HFA_134a propellant
  Arms: Foster 100/6mg pMDI

SUMMARY:
The purpose of this study is to demonstrate the non-inferiority of Foster 100/6mg NEXThaler versus Foster 100/6mg pMDI in terms of pulmonary function in asthmatic patients, as well as the effect of the test treatments in terms of additional lung function parameters and clinical outcome measures. The purpose is also to assess the safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients, Chinese ethnicity aged >18 years with a clinical diagnosis of asthma for a minimum of 6 months prior to visit 1 confirmed by a chest physician according to International guidelines updated 2016 Global Initiative Asthma (GINA).
* Positive Response to Reversibility Test.
* FEV 1 (Forced Expiratory Volume within the first second) >80% of the predicted normal value after appropriate washout from bronchodilators.
* Patients on previous regular treatment at a stable dose for at least 3 months prior to visit 1 with either high daily dose of ICS ( Inhaled Corticosteroids) or medium daily dose of ICS

Exclusion Criteria:

* Pregnant or lactating woment
* Intermittent asthma or asthma occurring only duting episodic exposure to an allergen or a chemical sensitizer
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) as defined by the current Glocal Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines updated 2016
* Current smokers, or ex-smokers
* Severe asthma exacerbation leading to intake of systemic corticosteroids (> 10 days) within 1 month prior to inclusion or moderate/severe asthma exacerbations
* Patients treated with monoclonal antibodies
* Patients treated with non-potassium sparing diuretics
* Patients treated with monoamine oxidase inhibitors and tricyclic antidepressants
* Patients who are receiving therapy that could interact with steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Demonstration of non-inferiority of Foster 100/6mg NEXThaler versus Foster 100/6mg pMDI in terms of pulmonary function | Baseline to week 12
  Change from Baseline to the entire treatment period in average pre-dose morning Peek Expiratory flow (PEF)

SECONDARY OUTCOMES:
Evaluation of the effect of the test treatment in terms of additional lung function parameters and clinical outcome measures, and assessement of the safety and tolerability | Baseline to week 12
  Changes in average pre-dose morning Peek Expiratory flow (PEF)
Evaluation of the effect of the test treatment in terms of additional lung function parameters and clinical outcome measures, and assessement of the safety and tolerability | Baseline to week 12
  Changes in average pre-dose evening PEF Daily PEF variability Average use fo rescue medication (number of puffs/day) Percentage of rescue-use free days Average total morning asthma symptom scores Average total evening asthma symptom scores Percentage of asthma symptoms-free days Percentage of asthma control days
Evaluation of the effect of the test treatment in terms of additional lung function parameters and clinical outcome measures, and assessement of the safety and tolerability | Baseline to Week 12
  Changes from Baseline in pre-dose morning Forced Expiratory Volume (FEV1) and Forced Vital Capacity (FVC) at each clinic visit.
Evaluation of the effect of the test treatment in terms of additional lung function parameters and clinical outcome measures, and assessement of the safety and tolerability | Baseline to week 12
  Change from Baseline to end of treatment in the Asthma Control Questionnaire (ACQ)

CONTACTS AND LOCATIONS:
Overall Officials: Jinping MD Zheng, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (51):
- China (51):
  - Chiesi Clinical Trial site 15641, Hefei, Anhui
  - Chiesi Clinical Trial site 15682, Beijing, Beijing Municipality
  - Chiesi Clinical Trial site 15663, Beijing, Beijing Municipality
  - Chiesi Clinical Trial site 15662, Foshan, Guangdong
  - Chiesi Clinical Trial site 15671, Guangzhou, Guangdong
  - Chiesi clinical Trial Site 15610, Guangzhou, Guangdong
  - Chiesi clinical Trial site 15656, Guangzhou, Guangdong
  - Chiesi Clinical Trial site 15668, Guangzhou, Guangdong
  - Chiesi Clinical Trial site 15677, Huizhou, Guangdong
  - Chiesi Clinical Trial site 15683, Shenzhen, Guangdong
  - Chiesi Clinical Trial site 15608, Shenzhen, Guangdong
  - Chiesi Clinical Trial site 15607, Zhanjiang, Guangdong
  - Chiesi Clinical Trial site 15610, Guangzhou, Guangzhou
  - Chiesi Clinical Trial site 15668, Guangzhou, Guangzhou
  - Chiesi Clinical Trial site 15673, Haikou, Hainan
  - Chiesi Clinical Trial site 15678, Qiqihar, Heilongjiang
  - Chiesi Clinical Trial site 15681, Xinxiang, Henan
  - Chiesi Clinical Trial site 15679, Zhengzhou, Henan
  - Chiesi Clinical Trial site 15614, Wuhan, Hubei
  - Chiesi Clinical Trial site 15661, Wuhan, Hubei
  - Chiesi Clinical Trial site 15675, Hengyang, Hunan
  - Chiesi Clinical Trial site 15643, Changzhou, Jiangsu
  - Chiesi Clinical Trial site 15674, Pingxiang, Jiangxi
  - Chiesi Clinical Trial site 15676, Jilin, Jilin
  - Chiesi clinical Trial site 15621, Shenyang, Liaoning
  - Chiesi clinical Trial site 15619, Nanchang, Nanchang
  - Chiesi Clinical Trial site 15650, Hohhot, Neimenggu
  - Chiesi clinical Trial site 15659, Hohhot, Neimenggu
  - Chiesi Clinical Trial site 15630, Shanghai, Shanghai Municipality
  - Chiesi Clinical Trial site 15664, Shanghai, Shanghai Municipality
  - Chiesi Clinical Trial site 15654, Shanghai, Shanghai Municipality
  - Chiesi Clinical Trial site 15631, Shanghai, Shanghai Municipality
  - Chiesi Clinical Trial site 15665, Shanghai, Shanghai Municipality
  - Chiesi Clinical Trial site 15625, Taiyuan, Shanxi
  - Chiesi Clinical Trial site 15611, Shijiazhuang, Shijiazhuang
  - Chiesi Clinical Trial site 15633, Chengdu, Sichuan
  - Chiesi Clinical Trial site 15680, Chongqing, Sichuan
  - Chiesi Clinical Trial site 15642, Tianjin, Tianjin Municipality
  - Chiesi Clinical Trial site 15634, Tianjin, Tianjin Municipality
  - Chiesi Clinical Trial site 15626, Xi'an, Xian
  - Chiesi Clinical Trial site 15672, Beijing
  - Chiesi clinical Trial site 15636, Beijing
  - Chiesi Clinical Trial site 15638, Chongqing
  - Chiesi Clinical Trial site 15670, Guizhou
  - Chiesi clinical Trial Site 15611, Hebei
  - Chiesi Clinical trial site 15660, Jilin
  - Chiesi Clinical Trial site 15628, Shanghai
  - Chiesi clinical trial site 15637, Shanghai
  - Chiesi Clinical Trial site 15666, Shenzhen
  - Chiesi clinical Trial site 15633, Sichuan
  - Chiesi Clinical Trial site 15669, Ürümqi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zheng J, Zhang J, Fu X, Lin C, Zhang X, Mei X, Corradi M, Cappellini G, Calabro E, Zhu C, Topole E. Comparison of extrafine beclomethasone dipropionate/formoterol fumarate dry powder inhaler and pressurized metered-dose inhaler in Chinese patients with asthma: the FORTUNE study. J Asthma. 2024 Apr;61(4):360-367. doi: 10.1080/02770903.2023.2272816. Epub 2023 Nov 1. PMID 37878325
- See also: Lay Summary of clinical trial results is available both in English and Chinese on the Chiesi Group web-site, along with a copy of the CSR synopsis. — https://www.chiesi.com/en/chiesi-clinical-study-register/